CLINICAL TRIAL: NCT06008470
Title: Investigation of Respiratory Muscle Strength, Exercise Capacity, Physical Activity and Sleep Quality Level in Individuals With Covid-19 Infection
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, research asistant, Kırıkkale University
Other Study IDs: Gurbuz04
Record Dates: First submitted 2023-08-21; First posted 2023-08-23 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Sleep Disorder; Respiratory Failure
MeSH Terms: conditions — COVID-19; Sleep Wake Disorders; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid-19: Inclusion Criteria:
  * Literacy,
  * To be between the ages of 18-45,
  * To study at Kırıkkale University Faculty of Health Sciences
  * Volunteering to participate in the research,
  Interventions: Other: observational tests
- control
  Interventions: Other: observational tests

INTERVENTIONS:
Other: observational tests — Respiratory Muscle Strength Measurement In our study, respiratory muscle strength will be measured using a portable, electronic mouth pressure measuring device (MEC Pocket Spiro MPM100, Belgium). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurement is one of the most commonly used non-invasive methods to evaluate respiratory muscles.
  6 Minute Walk Test (6MWT): It has been used to assess physical activity and functional capacity in many pulmonary rehabilitation programs for patients with chronic pulmonary disease and limited respiratory capacity

SUMMARY:
COVID-19 infection was identified in Wuhan, China at the end of 2019 and turned into a pandemic in a short time. In our country, the pandemic continues at full speed and patients are being treated in various clinical pictures. In its clinical classification, the World Health Organization (WHO) divides COVID-19 disease into four stages: mild symptomatic disease, pneumonia, severe pneumonia, acute respiratory distress syndrome (ARDS), sepsis and advanced stage with septic shock. Case reports and cross-sectional studies report a list of more than 200 different symptoms in the development of post COVID-19 syndrome. Shortness of breath, persistent smell and taste disturbances, fatigue and neuropsychological symptoms (headache, memory loss, slowed thinking, anxiety, depression and sleep disturbances) are the most commonly reported symptoms. Musculoskeletal symptoms such as pain (myalgia), muscle weakness, arthralgia and fatigue are also common. Exercise endurance tests are used to predict the prognosis of the disease in chronic lung diseases, to determine functional exercise capacity, to evaluate the response of the disease to treatment and to interpret the results of clinical trials. Covid-19-induced lung infections and long periods of isolation may have negative effects on respiratory muscle strength, pulmonary function values and physical activity level. It has been reported that only one week of bed rest can cause serious muscle loss of up to 20%. Covid-19 infection increases the likelihood of asthma-like symptoms. In some cases, pneumonia and increased dyspnea are also seen. When volleyball players with Covid-19 infection were examined, respiratory muscle strength and fev1/fvc values were lower than expected.

When looking at the interaction between infections and sleep, it was observed that different infections had different effects on sleep, with some infections increasing the amount of sleep while others decreased it. The increase in inflammatory mediators associated with systemic infection is thought to increase the amount of REM sleep and total sleep duration, perhaps in an effort to conserve energy and counteract infection. Some infections have a negative effect on the immune system, reducing the amount of sleep. Covid infection is also thought to have negative effects on sleep. The symptoms of COVID-19 in the chronic phase can further negatively affect physiological, psychological and social outcomes, physical activity and ultimately muscle performance and quality. Post-infection physical function and fitness can worsen even two years after the disease.

In COVID-19 patients recovering 3 months after hospital discharge, limitations were mainly related to reduced muscle mass, low oxidative capacity or both, rather than cardiac or respiratory exercise limitation.

Symptoms experienced during Covid-19 infection are thought to have negative effects on exercise endurance. In order to meet the metabolic needs of the musculoskeletal system muscles during exercise, cardiac output, ventilation, pulmonary and systemic blood flow, oxygen and carbon dioxide exchange in a way to maintain acid-base balance and oxygenation, and their compatible response to each other are required. Exercise endurance assessments are an important parameter to determine the functional level of the patient. Eighty-eight percent of individuals with Covid-19 infection showed a decrease in respiratory muscle strength in the evaluation performed 5 months later. The direct effect of respiratory muscles may cause permanent dyspnea problems. Muscle strength, exercise capacity, dyspnea perception, fatigue severity perception, pain, balance, kinesiophobia, psychosocial and cognitive status, quality of life should be routinely evaluated in the post-COVID-19 period in patients admitted to the clinic, and a targeted functional rehabilitation program should be prepared in the light of these evaluations, taking these parameters into consideration during the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* - Literacy,
* To be between the ages of 18-45,
* To study at Kırıkkale University Faculty of Health Sciences
* Volunteering to participate in the research,

Exclusion Criteria:

* - Individuals who are professional athletes with musculoskeletal system, cardiopulmonary system, metabolic system and other systemic problems that may affect physical activity habits will not be included in the study.
* A repeat COVID-19 PCR test positivity within the last 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As a result of the power analysis performed according to the sample article, it was calculated that 95% power would be obtained with 95% confidence when 30 people were included in each group for a total of 60 people. The MMP value was taken as the primary outcome measure. The impact factor was calculated as 0.958. Individuals will be selected from the students of our department. 30 people are post-covid, 30 people are healthy control group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT): | 6 min
  The 6DYT is a simple, low-cost test that monitors blood pressure (BP), heart rate (HR), respiratory frequency (RF), 'pulse' oxygen saturation (SpO2), score on the Borg Scale and distance walked. This test allows determination of physical fitness and VO2max and also assesses the patient's capacity and exercise tolerance.

SECONDARY OUTCOMES:
Sleep Quality Level(pitsburg sleep scale) | 5 minute
  The PSQI was developed by Buysse et al. (1989) and adapted into Turkish by Ağargün et al. (1996). The PSQI is a 19-item self-report scale that evaluates sleep quality and disturbance in the past one month. It consists of 24 questions, 19 questions are self-report questions and 5 questions are questions to be answered by a spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficacy, Sleep Disorder, Sleep Medication Use and Daytime Dysfunction. Each component is evaluated on a 0-3 point scale. The total score of the 7 components gives the total scale score. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality"
Respiratory Muscle Strength Measurement | 10 min
  In our study, respiratory muscle strength will be measured using a portable, electronic mouth pressure measuring device (MEC Pocket Spiro MPM100, Belgium). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurement is one of the most commonly used non-invasive methods to evaluate respiratory muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided